CLINICAL TRIAL: NCT00553189
Title: A Phase I Study of ABT-888 in Combination With Topotecan Hydrochloride in Adults With Refractory Solid Tumors and Lymphomas
Brief Title: Safety Study of ABT-888 Plus Topotecan Hydrochloride to Treat Patients With Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 070203; 07-C-0203; NCT01445353 (obsolete NCT alias)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-28

CONDITIONS: Solid Tumors; Lymphomas
Keywords: PARP Inhibitor; Advanced Cancer; Combination Therapy; Early Trial; DNA Damage Repair; Topotecan; Cancer; Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — veliparib; Topotecan

INTERVENTIONS:
Drug: ABT-888
Drug: Topotecan

SUMMARY:
Background:

* PARP is an enzyme that is involved in the repair of damage to DNA. Levels of the enzyme are higher in tumor cells than in normal cells, and may play a part in resistance to cancer chemotherapy and radiation therapy. ABT-888 is an experimental drug that inhibits PARP and may help to increase the effectiveness of cancer treatments designed to damage DNA in cancer cells.
* Topotecan is a drug approved by the Food and Drug Administration for treating certain cancers.
* This dose escalation study will test the two drugs at successively higher doses in small groups of patients until the highest safe dose is determined.

Objectives:

* To test the safety of the combination of ABT-888 and Topotecan (TPT) and determine the highest dose of each drug that can be safely given to humans. This is the maximum tolerated dose (MTD).
* To learn how the combination of ABT-888 and TPT works in humans and how the body handles the drugs.
* To determine the side effects of the combination of ABT-888 and TPT at the tested doses.

Eligibility:

-Patients with solid tumors, lymphomas and chronic lymphocytic leukemia whose disease has progressed following standard therapy or for whom standard treatments are not available.

Design:

* ABT-888 and TPT are given in 21-day treatment cycles. At the start of the study, TPT is infused through a vein over 30 minutes about a week before cycle 1 starts. Starting on day 1 of cycle 1, ABT-888 is given by mouth twice a day for 7 days. TPT is given through a vein daily for 4 days starting on day 2. After the last dose of ABT-888 day 7, no more treatment is given for the rest of the 21-day cycle.
* For the remaining cycles, ABT-888 is given twice a day by mouth on days 1 to 7 of each cycle, and TPT is given through a vein daily on days 1 to 5 of each cycle.
* The first three to six patients enrolled in the study take the smallest study dose of the drugs. If they do not develop significant adverse side effects, successive small groups of patients take the drug at increasingly higher doses until the MTD is reached. Additional patients enrolled receive the MTD.
* Patients have periodic clinic visits for their TPT infusions and for tests and examinations. Evaluations include measurement of vital signs, physical examinations, blood and urine tests, electrocardiograms and CT or other imaging tests, such as ultrasound or MRI. Tumor biopsies may be requested to study the effects of the drugs on the...

DETAILED DESCRIPTION:
Background:

* The PARP family of enzymes is characterized by the ability to poly (ADP-ribosyl)ate protein substrates. PARP-1 and PARP-2 play a critical role in the maintenance of genomic stability by regulating a variety of DNA repair mechanisms.
* Poly (ADP-ribosylated) PARP-1 has been shown to block the formation of topo 1-DNA cleavage and accelerate the removal of camptothecin-stabilized topo 1-DNA complexes. PARP-1 inhibition may therefore prevent efficient repair of DNA damage induced by topoisomerase 1 inhibitors. ABT-888 is an oral PARP inhibitor and topotecan is a topoisomerase I inhibitor.

Objectives:

* Establish the safety and tolerability of the combination of ABT-888 with topotecan hydrochloride in patients with refractory solid tumors and lymphomas.
* Establish the maximum tolerated dose of the combination of ABT-888 with topotecan hydrochloride.
* Evaluate the pharmacokinetics of each agent alone and in combination.
* Determine the effects of the study treatment on the level of PARP inhibition and DNA damage in PBMCs and tumor samples.

Eligibility:

* Patients with histologically documented solid tumors and lymphoid malignancies (lymphoma and CLL) whose disease has progressed following standard therapy or who have no acceptable standard treatment options.
* No major surgery, radiation or chemotherapy within four weeks prior to study enrollment, and recovered from toxicities of prior therapies to at least eligibility levels.

Study Design:

* Cycle 1, dose levels -1 to 7 and 1B: Topotecan (TPT) will be administered intravenously over 30 minutes as a single dose on days 1-5. Starting on day 2, ABT-888 will be administered orally twice a day on a q12 hour schedule for 4 days (D2-5). Following the completion of study drug administration on day 5, no further treatment will be administered for the rest of this 21-day cycle. Growth factors will be administered prophylactically starting Cycle 1 to patients on dose level 1B only.
* Cycle 2 and beyond, dose levels -1 to 7 and 1B: ABT-888 will be administered twice a day on a q12 hour schedule orally on days 1-5. TPT will be given IV daily from days 1-5, in a 21-day cycle. Growth factors will be administered prophylactically to patients on dose level 1B only.
* All cycles, dose levels -2 and 1A to 5A: ABT-888 will be administered on day 1 only for dose levels -2 and 1A, 2A, 3A, and 4A. For dose level 5A, ABT-888 will be administered on days 1 and 2 of each cycle. TPT will be given IV daily from days 1-5, in a 21-day cycle.
* Dose escalation will proceed as outlined below. Once maximum tolerated dose (MTD) is established, 6 additional patients will be enrolled at the MTD to further define the dose and evaluate PD studies at this dose level.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients with histologically documented solid tumors and lymphoid malignancies (lymphoma and CLL) who are refractory to standard therapy or who have no acceptable standard treatment options. Patients with lymphoid malignancies will be eligible if their disease has progressed following standard therapy and if stem cell transplantation is not indicated or has been refused.
2. Any prior therapy must have been completed greater than or equal to 4 weeks prior to enrollment on protocol and the participant must have recovered to eligibility levels (CTCAE Grade less than or equal to 1) from prior toxicity. Prior radiation or surgery should have been completed greater than or equal to 4 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study, and should have recovered to eligibility levels from any toxicities.
3. Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of ABT-888 in patients less than 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase I combination trials.
4. ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60 percent).
5. Life expectancy of greater than 3 months.
6. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count greater than or equal to 1,500/mcL
   * platelets greater than or equal to 100,000/mcL
   * total bilirubin less than 1.5 times institutional upper limit of normal
   * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal
   * creatinine less than 1.5 times institutional upper limit of normal

   OR

   -creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels above institutional normal.
7. The effects of ABT-888 on the developing human fetus are unknown. For this reason and because topotecan hydrochloride used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after completion of study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study, and should have recovered to eligibility levels from any toxicities.

   Patients who have been administered ABT-888 as part of a single or limited dosing study, such as a Phase 0 study, should not be excluded from participating in this study solely because of receiving prior ABT-888.

   Patients who have received prior TPT should not be excluded solely because of receiving prior TPT.
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, prolonged QTc interval (greater than msec), or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with known brain mestastases or a history of seizures are excluded from this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-08-09; Primary Completion 2008-02-01 (Actual); Study Completion 2011-09-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the combination of ABT-888 with topotecan hydrochloride in patients with refractory solid tumors and lymphomas; Establish the maximum tolerated dose of ABT-888 with topotecan hydrochloride.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetic of each agent alone and in combination; determine the effects of the study treatment on the level of PARP inhibition and DNA damage in PBMCs and tumor samples.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ame JC, Rolli V, Schreiber V, Niedergang C, Apiou F, Decker P, Muller S, Hoger T, Menissier-de Murcia J, de Murcia G. PARP-2, A novel mammalian DNA damage-dependent poly(ADP-ribose) polymerase. J Biol Chem. 1999 Jun 18;274(25):17860-8. doi: 10.1074/jbc.274.25.17860. PMID 10364231
- [Background] Ame JC, Spenlehauer C, de Murcia G. The PARP superfamily. Bioessays. 2004 Aug;26(8):882-93. doi: 10.1002/bies.20085. PMID 15273990
- [Background] Berger NA, Adams JW, Sikorski GW, Petzold SJ, Shearer WT. Synthesis of DNA and poly(adenosine diphosphate ribose) in normal and chronic lymphocytic leukemia lymphocytes. J Clin Invest. 1978 Jul;62(1):111-8. doi: 10.1172/JCI109094. PMID 659624
- [Derived] Kummar S, Chen A, Ji J, Zhang Y, Reid JM, Ames M, Jia L, Weil M, Speranza G, Murgo AJ, Kinders R, Wang L, Parchment RE, Carter J, Stotler H, Rubinstein L, Hollingshead M, Melillo G, Pommier Y, Bonner W, Tomaszewski JE, Doroshow JH. Phase I study of PARP inhibitor ABT-888 in combination with topotecan in adults with refractory solid tumors and lymphomas. Cancer Res. 2011 Sep 1;71(17):5626-34. doi: 10.1158/0008-5472.CAN-11-1227. Epub 2011 Jul 27. PMID 21795476